CLINICAL TRIAL: NCT03177161
Title: Assessment of Patient Reported Health Status Questions Via Four Different Methods of Administration, in Stroke Survivors. A Randomised Controlled Trial. A Non-inferiority Study of the Response Rate for Four Alternative Methods of Administration of 15 Patient Reported Health Status Questions in Stroke Survivors.
Brief Title: Assessment of Patient Reported Health Status Questions Via Four Different Methods of Administration, in Stroke Survivors.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Jonathan Hewitt (Other)
Collaborators: Stroke Implementation Group (Wales) (Unknown)
Responsible Party: Sponsor-Investigator, Dr Jonathan Hewitt, Clinical Senior Lecturer (Cardiff University) & Honorary Consultant Physician (ABUHB), Aneurin Bevan University Health Board
Organization: Aneurin Bevan University Health Board (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRAS 222226
Record Dates: First submitted 2017-05-26; First posted 2017-06-06 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Stroke; Cerebral Infarction; Cerebral Hemorrhage; Stroke Hemorrhagic; Stroke, Ischemic; Stroke of Uncertain Pathology
Keywords: PROM; Patient Reported Outcome Measure; PROMIS; PROMIS-10; PROMIS Global Health; RiksStroke; ICHOM; International Consortium for Health Outcomes Measurement; Wales; Administration; Method; Delivery
MeSH Terms: conditions — Stroke; Cerebral Infarction; Cerebral Hemorrhage; Hemorrhagic Stroke; Ischemic Stroke

STUDY DESIGN:
Masking Description: Participants will not be made aware of the other modes of delivery available and will be assigned a single method of delivery prior to consent.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Postal Questionnaire (Experimental)
  Interventions: Other: 15 Patient Reported Health Status Questions
- Online Questionnaire (Experimental)
  Interventions: Other: 15 Patient Reported Health Status Questions
- Face-to-face Questionnaire (Experimental)
  Interventions: Other: 15 Patient Reported Health Status Questions
- Telephone Questionnaire (Experimental)
  Interventions: Other: 15 Patient Reported Health Status Questions

INTERVENTIONS:
Other: 15 Patient Reported Health Status Questions — The PROMIS-10 Global Health, three single item questions (ambulation, toileting, and dressing) that have been borrowed from the RiksStroke (The National Quality Register for Stroke - Sweden) and two further questions on feeding and communication have been included from the ICHOM Standard Set for Stroke.

SUMMARY:
A Patient Reported Outcome Measure (PROM) is a questionnaire that asks patients for their views on their own health or the impact of healthcare they have received on their health and quality of life (RCN, 2011). The benefit of PROMS is that they gather information from the patient's perspective, which offers great potential to improve the quality and outcomes of health services (Department of Health 2011).

There is a PROM (the PROMIS-10 Global Health) and a number of extra questions that are recommended for use in people who have had a stroke by the International Consortium for Health Outcomes Measurement, but the best way of delivering these questions for stroke survivors is unknown.

At present, the NHS in England, Scotland and Wales are required to offer every stroke survivors a 6 month post stroke follow-up appointment. Currently, the information collected at the 6 month review is not from the patient's perspective and the best method of collecting this information has not been established. The Sentinel Stroke National Audit Programme (SSNAP) which is led by the Royal College of Physicians in London promote the 6 month follow-up assessment. SSNAP recognise that currently 4 different methods of 6 month follow-up appointment occur. The current methods in use are face-to-face assessment, telephone interview, online questionnaire or postal questionnaire.

The aim of this research is to understand if there is a difference between these 4 methods of delivering these questions in people who have had a stroke.

As part of the 6 month review this research study will assess the response rate for 15 Patient Reported Health Status questions across the 4 recognised methods of delivery;

* Face-to-Face
* Telephone
* Online
* Post

To conduct this research study a sample of 808 stroke survivors will be asked to take part in the research. From these 808 people, 202 participants will be randomly assigned to each method of administration (Face-to-Face Interview, Telephone Interview, Postal Questionnaire and Online Questionnaire).

The questionnaires received by the research team will not record any personally identifiable information. The data will then be utilised by the researchers for statistical analysis in order to identify, which method of the 4 methods of administration, under investigation, is the most acceptable for stroke survivors. The conclusions of this research will inform the roll-out of the most appropriate method of delivering the 6 month stroke follow-up review for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of stroke either Cerebral Infarct (ICD I63), Cerebrovascular Haemorrhage (ICD161) or Stroke, not specified as haemorrhage or infarction (ICD I64).
* Patients over 18 years old (≥ 18 years old)
* Had a diagnosis of stroke within the last 4-8 months (Stroke diagnosis ≥ 4months to ≤ 8 months)

Exclusion Criteria:

* Diagnosis of a Transient Ischaemic Attack (ICD G45)
* Diagnosis of a Subarachnoid Haemorrhage (ICD I60)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2017-08-12 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Total response rate for all 4 methods of delivery | 120 to 240 days post index event
  As defined by response rate. This will be measured by the number of individuals that return the questionnaire for each of the four allocation groups.

SECONDARY OUTCOMES:
Total response rate across the four different methods of administration for 15 Patient Reported Health Status questions with people with communication issues (e.g. aphasia) | 120 to 240 days post index event
Total response rate across the four different methods of administration for 15 Patient Reported Health Status questions by stroke severity (as defined by NIHSS on admission) | 120 to 240 days post index event
Total response rate across the four different methods of administration for 15 Patient Reported Health Status questions by stroke type (as defined by ICD classification) | 120 to 240 days post index event

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Hewitt, MBBS, FRCP (Glas), MSc, PhD, Study Director — Cardiff University & Aneurin Bevan University Health Board
Locations (4):
- United Kingdom (4):
  - Ysbyty Ystrad Fawr, Ystrad Mynach, Caerphilly
  - Royal Gwent Hospital, Newport, Gwent
  - Nevill Hall Hospital, Abergavenny, Monmouthshire
  - Prince Charles Hospital, Merthyr Tydfil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith A, Pennington A, Carter B, Gething S, Price M, White J, Dewar R, Hewitt J. Acceptability of the method of administration of a patient-reported outcome measure (PROM) with stroke survivors, a randomised controlled trial protocol. Trials. 2018 Jul 3;19(1):349. doi: 10.1186/s13063-018-2694-4. PMID 29970156
- [Derived] Hewitt J, Pennington A, Smith A, Gething S, Price M, White J, Dewar R, Carter B. A multi-centre, UK-based, non-inferiority randomised controlled trial of 4 follow-up assessment methods in stroke survivors. BMC Med. 2019 Jul 2;17(1):111. doi: 10.1186/s12916-019-1350-5. PMID 31262317